CLINICAL TRIAL: NCT03987932
Title: NEAT!2 Sedentary Behavior Reduction Intervention for Individuals With Past or Present Knee Symptoms, Injuries, or Surgeries
Brief Title: NEAT!2 Sedentary Behavior Reduction for Individuals With Past or Present Knee Symptoms, Injuries, or Surgeries
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Christine A Pellegrini, PhD, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00085868
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Results first posted 2021-06-22 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Sedentary Lifestyle; Knee Osteoarthritis; Knee Injuries; Knee Pain Chronic
MeSH Terms: conditions — Sedentary Behavior; Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NEAT!2 (Experimental): Participants will be asked to use the NEAT!2 app for 3 months after randomization. App use between 4-6 months is optional.
  Interventions: Behavioral: NEAT!2
- NEAT!2+Calls (Experimental): Participants will be asked to use the NEAT!2 app for 3 months after randomization. In addition, participants will receive bi-weekly coaching calls over 3 months. App use between 4-6 months is optional.
  Interventions: Behavioral: NEAT!2+Calls
- Delayed NEAT!2 (Other): Participants will receive the NEAT!2 app to use between 3 and 6 months.
  Interventions: Behavioral: Delayed NEAT!2

INTERVENTIONS:
Behavioral: NEAT!2 — Participants randomized to NEAT!2 will have their NEAT!2 app turned on after randomization. When 30 minutes of continuous non-movement or sedentary time is detected, the NEAT!2 app will provide a vibration or audio notification as well as display a reminder on the phone's lock/home screen. Participants will be asked to use the app for the 3 months of the intervention. Participants will be given an initial goal to reduce total sedentary time by 30 minutes/day, ultimately progressing to a 90 minute/day reduction by 3 months. After the 3-month assessment, participants randomized to NEAT!2 will have the option to continue using the app until 6 months.
  Arms: NEAT!2
Behavioral: NEAT!2+Calls — Participants in this group will have their NEAT!2 app turned on after randomization. In addition, to receiving the identical app and given the same goals as participants randomized to NEAT!2, NEAT!2+Calls participants will receive 10-15 minute bi-weekly coaching calls. After the 3-month assessment, participants will have the option to continue using the app until 6 months. During this time, participants will not receive any coaching calls.
  Arms: NEAT!2+Calls
Behavioral: Delayed NEAT!2 — Participants randomized to Delayed NEAT!2 will not receive any contact or app between baseline and 3 months. However, after completing the 3-month assessment, participants will receive the NEAT!2 application. Participants will then have the option to use the app between 3 and 6 months.
  Arms: Delayed NEAT!2

SUMMARY:
This study will evaluate the effectiveness of an mHealth sedentary reduction program over a 6-month period of time in adults with past or present knee symptoms, injuries, or surgeries.

DETAILED DESCRIPTION:
Sedentary behavior, in excess, is associated with numerous health consequences including poor physical function. Older adults with symptomatic knee pain spend the majority of their waking hours engaging in sedentary behaviors. To reduce the risk of disability, improve quality of life, and prevent deterioration in physical function, it is imperative the investigators develop ways to reduce sedentary time. Smartphone ownership among older adults is increasing and may provide a scalable opportunity to disseminate a sedentary reduction intervention. Therefore, this study aims to evaluate and compare changes in sedentary behavior and physical function between an mHealth sedentary reduction, mHealth intervention plus coaching, and delayed mHealth group. Sedentary behavior and physical function will be assessed at baseline, 1 month, 3 months, and 6 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 40 years of age
* Own an Android or Apple smartphone
* Have their smartphone near them (in their pocket, in their hand, or within 10 feet of them) for >50% of their waking day
* Be willing to download the study application and be compatible on their smartphone
* Spend at least 7 hours/day sitting
* Have at least 4 days of valid accelerometer data at baseline
* Have knee pain (at least one knee with pain, aching, or stiffness on most days for one month of the last 12 months), knee injury, or knee replacement within the last 5 years
* Read, speak, and understand English

Exclusion Criteria:

* Have any contraindications to activity
* Have a mobility limiting comorbidity
* Have a scheduled surgery within the next 6 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-06-22 (Actual); Primary Completion 2020-09-09 (Actual); Study Completion 2020-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NEAT!2 | NEAT!2+Calls | Delayed NEAT!2
Started (Study stopped due to COVID-19) | 4 | 3 | 4
1 Month | 4 | 2 | 3
3 Months | 4 | 2 | 3
6 Months | 2 | 2 | 2
Completed (Study stopped due to COVID-19) | 2 | 2 | 2
Not Completed | 2 | 1 | 2
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Non-study related elective surgery | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NEAT!2 | NEAT!2+Calls | Delayed NEAT!2 | Total
Number analyzed (Participants) | 4 | 3 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 3 | 9
  >=65 years | 0 | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (10.2) | 60.2 (6.9) | 48.8 (9.0) | 55.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 2 | 1 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 3 | 4 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 4 | 11
Timed Up and Go [Mean (Standard Deviation); unit: seconds] | 7.2 (0.3) | 6.5 (1.1) | 8.3 (3.7) | 7.4 (2.2)
Six Minute Walk [Mean (Standard Deviation); unit: feet] | 1491.2 (226.7) | 1553.1 (223.3) | 1496.8 (476.0) | 1510.1 (306.8)
Chair Stands [Mean (Standard Deviation); unit: chair stands] | 9.3 (2.5) | 12.0 (3.6) | 10.0 (4.5) | 10.3 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sedentary Behavior at 1 Month
Description: Daily sedentary behavior objectively measured by activpal
Time Frame: Baseline to 1 month
Measure: Mean (Standard Deviation); unit: change in minutes
Arm/Group | NEAT!2 | NEAT!2+Calls | Delayed NEAT!2
Number analyzed (Participants) | 4 | 2 | 4
change in minutes | -33.7 (119.2) | -24.5 (23.0) | 32.0 (44.2)

2. Primary Outcome: Change in Sedentary Behavior at 3 Months
Description: Daily sedentary behavior objectively measured by activpal
Time Frame: Baseline to 3 months
Measure: Mean (Standard Deviation); unit: change in minutes
Arm/Group | NEAT!2 | NEAT!2+Calls | Delayed NEAT!2
Number analyzed (Participants) | 4 | 2 | 3
change in minutes | 43.4 (99.1) | -44.7 (39.4) | 12.9 (14.3)

3. Secondary Outcome: Change in Timed Up & Go at 1 Month
Description: Physical function assessed by Timed Up & Go (seconds)
Time Frame: Baseline to 1 month
Population: Data collection for function tests stopped after COVID-19
Measure: Mean (Standard Deviation); unit: change in seconds
Arm/Group | NEAT!2 | NEAT!2+Calls | Delayed NEAT!2
Number analyzed (Participants) | 3 | 2 | 3
change in seconds | -.4 (1.0) | -.4 (1.5) | -.1 (1.0)

4. Secondary Outcome: Change in Chair Stands at 1 Month
Description: Physical function assessed by Chair Stand Test (# stands in 30 seconds)
Time Frame: Baseline to 1 month
Population: Data collection for function tests stopped after COVID-19
Measure: Mean (Standard Deviation); unit: change in chair stands
Arm/Group | NEAT!2 | NEAT!2+Calls | Delayed NEAT!2
Number analyzed (Participants) | 3 | 2 | 3
change in chair stands | .3 (1.2) | 2 (1.4) | .3 (1.2)

5. Secondary Outcome: Change in 6 Minute Walk at 1 Month
Description: Physical function assessed by 6 minute walk (total feet)
Time Frame: Baseline to 1 month
Population: Data collection for function tests stopped after COVID-19
Measure: Mean (Standard Deviation); unit: change in feet
Arm/Group | NEAT!2 | NEAT!2+Calls | Delayed NEAT!2
Number analyzed (Participants) | 3 | 2 | 3
change in feet | 76.0 (130.7) | 74 (104.7) | 89.0 (123.1)

6. Secondary Outcome: Change in Timed Up & Go at 3 Months
Description: Physical function assessed by Timed Up & Go (seconds)
Time Frame: Baseline to 3 months
Population: Data collection for function tests stopped after COVID-19
Measure: Mean (Standard Deviation); unit: change in seconds
Arm/Group | NEAT!2 | NEAT!2+Calls | Delayed NEAT!2
Number analyzed (Participants) | 3 | 2 | 3
change in seconds | -.3 (1.4) | -1.1 (1.0) | -.6 (.7)

7. Secondary Outcome: Change in Chair Stands at 3 Months
Description: Physical function assessed by Chair Stand Test (# stands in 30 seconds)
Time Frame: Baseline to 3 months
Population: Data collection for function tests stopped after COVID-19
Measure: Mean (Standard Deviation); unit: change in chair stands
Arm/Group | NEAT!2 | NEAT!2+Calls | Delayed NEAT!2
Number analyzed (Participants) | 3 | 2 | 3
change in chair stands | 2.3 (.6) | 3.0 (2.8) | -.7 (2.9)

8. Secondary Outcome: Change in 6 Minute Walk at 3 Months
Description: Physical function assessed by 6 minute walk (total feet)
Time Frame: Baseline to 3 months
Population: Data collection for function tests stopped after COVID-19
Measure: Mean (Standard Deviation); unit: change in feet
Arm/Group | NEAT!2 | NEAT!2+Calls | Delayed NEAT!2
Number analyzed (Participants) | 3 | 2 | 3
change in feet | 15.5 (11.4) | 678.2 (525.8) | 75.1 (81.9)

9. Other Pre Specified Outcome: Maintenance of Changes in Sedentary Behavior at 6 Months
Description: Daily sedentary behavior objectively measured by activpal
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: change in minutes
Arm/Group | NEAT!2 | NEAT!2+Calls | Delayed NEAT!2
Number analyzed (Participants) | 3 | 2 | 2
change in minutes | -30.5 (90.9) | -84.4 (138.3) | 80.2 (10.8)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | NEAT!2 | NEAT!2+Calls | Delayed NEAT!2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03987932/Prot_SAP_000.pdf